CLINICAL TRIAL: NCT03207256
Title: An Open Label Extension Trial of Ublituximab and/or Umbralisib (TGR-1202) in Combination With Other Novel Agents or as Single Agents in Subjects Currently Receiving Treatment on a TG Therapeutics Study.
Brief Title: Extension Trial of Ublituximab and TGR-1202 in Combination or as Single Agents in Subjects Currently Receiving Treatment on Ublituximab and/or TGR-1202 Trials
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTX-TGR-501
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Chronic Lymphocytic Leukemia; Non Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — umbralisib; ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TGR-1202 (Experimental): Oral TGR-1202 Daily
  Interventions: Drug: TGR-1202
- TGR-1202 + Ublituximab (Experimental): Oral TGR-1202 in combination with Ublituximab intravenous administration
  Interventions: Drug: TGR-1202 + Ublituximab

INTERVENTIONS:
Drug: TGR-1202 — Oral Daily TGR-1202
  Arms: TGR-1202
Drug: TGR-1202 + Ublituximab — Oral Daily TGR-1202 + Ublituximab IV Administration
  Arms: TGR-1202 + Ublituximab

SUMMARY:
This is an open label compassionate use trial of Ublituximab and TGR-1202 in combination or as single agents in patients currently receiving treatment on Ublituximab and/or TGR-1202 trials with B-cell Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be currently receiving treatment with ublituximab and/or TGR-1202 on a previously approved protocol.
* Subjects must have completed at least 6 cycles of therapy on their current protocol.

Exclusion Criteria:

* Subject progressed while receiving therapy with ublituximab and/or TGR-1202 while participating in their immediate previous trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Adverse Events of TGR-1202 and/or TGR-1202 + ublituximab treatment, including delayed toxicities | Evaluated at each planned visit through study completion, an average of 2 years
  Toxicity according to the investigator (Adverse events with NCI-CTC 4.0)

SECONDARY OUTCOMES:
Progression-free survival of TGR-1202 and/or TGR-1202 + ublituximab treatment | Evaluated at each planned visit through study completion, an average of 2 years
  Date of progression reported for each patient

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Tucson, Arizona
  - TG Therapeutics Investigational Trial Site, Fayetteville, Arkansas
  - TG Therapeutics Investigational Trial Site, Duarte, California
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, Atlanta, Georgia
  - TG Therapeutics Investigational Trial Site, Fort Wayne, Indiana
  - TG Therapeutics Investigational Trial Site, Coon Rapids, Minnesota
  - TG Therapeutics Investigational Trial Site, Omaha, Nebraska
  - TG Therapeutics Investigational Trial Site, Durham, North Carolina
  - TG Therapeutics Investigational Site, Canton, Ohio
  - TG Therapeutics Investigational Trial Site, Cincinnati, Ohio
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Denton, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Seattle, Washington
  - TG Therapeutics Investigational Trial Site, Milwaukee, Wisconsin